CLINICAL TRIAL: NCT01738620
Title: Quality of Life After Esophagectomy for Cancer - QOLEC1
Brief Title: Quality of Life After Esophagectomy for Cancer - Step 1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In October 2015 ICU's setting completely changed from an open concept 8-beds unit to a single bed isolated room.
Sponsor: University of Padova (Other)
Collaborators: Fondazione Guido Berlucchi (Other); Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: QOLEC1 - step 1
Record Dates: First submitted 2012-10-20; First posted 2012-11-30 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Esophageal Cancer; Sleep Disturbance; Quality of Life
Keywords: esophageal cancer; sleep disturbance; quality of life
MeSH Terms: conditions — Esophageal Neoplasms; Parasomnias | interventions — Intensive Care Units

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- psychological counseling+prevention of sleep disorders in ICU (Experimental): patients will receive both psychological counseling and interventions to prevent sleep disorders during their ICU stay
  Interventions: Behavioral: psychological counseling; Behavioral: prevention of sleep disorders in ICU
- psychological counseling (Experimental): patients will receive psychological counseling
  Interventions: Behavioral: psychological counseling
- prevention of sleep disorders in ICU (Experimental): interventions to prevent sleep disorders during their ICU stay
  Interventions: Behavioral: prevention of sleep disorders in ICU
- standard care (No Intervention): patients will receive standard care

INTERVENTIONS:
Behavioral: psychological counseling
  Arms: psychological counseling; psychological counseling+prevention of sleep disorders in ICU
Behavioral: prevention of sleep disorders in ICU
  Arms: prevention of sleep disorders in ICU; psychological counseling+prevention of sleep disorders in ICU

SUMMARY:
Background: A recent systematic review showed that patients undergoing esophagectomy for cancer had scores of physical function, vitality and performance of health in general significantly lower than those obtained from the reference population. The analysis of the quality of life at six months follow-up showed that the total score and physical function were better before surgery and symptoms-based scales indicated that the fatigue, dyspnoea and diarrhea were worse six months after esophagectomy. The objective of this study is therefore to assess the impact of esophageal resections for cancer on the quality of life of patients and to improve it through simple interventions of post operative care.

The study is divided into two steps.

This is step 1.

Patients will be randomized into four groups receiving respectively: psychological counseling for support plus appropriate measures to reduce sleep-wake rhythm disorders during ICU stay; psychological counseling alone; appropriate measures to reduce sleep-wake rhythm disorders during ICU stay alone; or standard care. The primary end point are the items SL (sleep disorder) and QL2 of the QLQ C30, and the secondary end point is the score of the PSQI.

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years old
* scheduled for esophagectomy for cancer

Exclusion Criteria:

* age below 18 years old
* incapability to autonomously fill in questionnaires
* primary language not italian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
items SL (sleep disorder) and QL2 of the QLQ C30 | 14 days (average time to hospital discharge)

SECONDARY OUTCOMES:
PSQI score | 14 days (average time to hospital discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Castoro, MD, Principal Investigator — Istituto Oncologico Veneto (IOV-IRCCS)
Locations (1):
- Istituto Oncologico Veneto (IOV-IRCCS), Padua, Padova, Italy

REFERENCES:
- [Derived] Geense WW, van den Boogaard M, van der Hoeven JG, Vermeulen H, Hannink G, Zegers M. Nonpharmacologic Interventions to Prevent or Mitigate Adverse Long-Term Outcomes Among ICU Survivors: A Systematic Review and Meta-Analysis. Crit Care Med. 2019 Nov;47(11):1607-1618. doi: 10.1097/CCM.0000000000003974. PMID 31464769
- [Derived] Scarpa M, Pinto E, Saraceni E, Cavallin F, Parotto M, Alfieri R, Nardi MT, Marchi MR, Cagol M, Castoro C; QOLEC Group. Randomized clinical trial of psychological support and sleep adjuvant measures for postoperative sleep disturbance in patients undergoing oesophagectomy. Br J Surg. 2017 Sep;104(10):1307-1314. doi: 10.1002/bjs.10609. Epub 2017 Jul 14. PMID 28707741